CLINICAL TRIAL: NCT07290881
Title: A Prospective Randomized Study Comparing the Postoperative Analgesic Efficacy of Anterior Iliac Block and Ilioinguinal-iliohypogastric Block in Inguinal Hernia Surgery
Brief Title: Comparing the Postoperative Analgesic Efficacy of Anterior Iliac Block and Ilioinguinal-iliohypogastric Block in Inguinal Hernia Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, ABDULHAKİM ŞENGEL, SPECİALİST, MD, ANESTHESİOLOGY AND REANİMATİON, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anterior iliac block
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group who underwent anterior iliac block (Active Comparator): In this patient group, an anterior iliac block will be administered in the postoperative period, and postoperative pain at the surgical site will be assessed.
  Interventions: Other: Patient group who underwent anterior iliac block
- Patient group who underwent ilioinguinal-iliohypogastric block (Active Comparator): In this patient group, an ilioinguinal-iliohypogastric block will be administered in the postoperative period, and postoperative pain at the surgical site will be assessed.
  Interventions: Other: Patient group who underwent ilioinguinal/iliohypogastric block

INTERVENTIONS:
Other: Patient group who underwent ilioinguinal/iliohypogastric block — Patient group who underwent ilioinguinal/iliohypogastric block
  Arms: Patient group who underwent ilioinguinal-iliohypogastric block
Other: Patient group who underwent anterior iliac block — Patient group who underwent anterior iliac block
  Arms: Patient group who underwent anterior iliac block

SUMMARY:
The primary aim of this study is to compare two postoperative analgesia techniques used in patients undergoing inguinal hernia surgery-(1) the anterior iliac block and (2) the ilioinguinal/iliohypogastric block-in terms of postoperative analgesia duration and patient satisfaction.

Effective postoperative analgesia in inguinal hernia surgery is crucial for improving patient comfort and reducing opioid consumption. Although ilioinguinal and iliohypogastric nerve blocks are commonly used for this purpose, their relatively limited dermatomal coverage may result in inadequate analgesia in some cases. The recently described Anterior Iliac Block has been proposed as an alternative to conventional techniques, offering potentially wider neural spread and more effective postoperative pain control. However, the efficacy and safety of this novel block have not yet been sufficiently evaluated in the literature.

DETAILED DESCRIPTION:
The primary aim of this study is to compare two postoperative analgesia techniques used in patients undergoing inguinal hernia surgery-(1) the anterior iliac block and (2) the ilioinguinal/iliohypogastric block-in terms of postoperative analgesia duration and patient satisfaction.

Effective postoperative analgesia in inguinal hernia surgery is crucial for improving patient comfort and reducing opioid consumption. Although ilioinguinal and iliohypogastric nerve blocks are commonly used for this purpose, their relatively limited dermatomal coverage may result in inadequate analgesia in some cases. The recently described anterior iliac block has been proposed as an alternative to conventional techniques, offering potentially wider neural spread and more effective postoperative pain control. However, the efficacy and safety of this novel block have not yet been sufficiently evaluated in the literature.

This study aims to compare the anterior iliac block with the ilioinguinal/iliohypogastric block in terms of postoperative pain control and patient satisfaction. The objective is to determine whether the anterior iliac block, through its broader dermatomal distribution, provides lower NRS pain scores, reduced analgesic requirements, and higher patient satisfaction compared with traditional nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* It includes patients aged 18-65 years
* Classified as ASA I-II
* Who are undergoing elective inguinal hernia surgery

Exclusion Criteria:

* Patients who did not wish to participate voluntarily
* Those with contraindications to the anterior iliac block or the Ilioinguinal/Iliohypogastric block,
* Pregnant or breastfeeding women
* Patients classified as ASA III-IV-V

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Akut ağrı (Sayısal Derecelendirme Ölçeği-NRS) | 0-1-3-6-12-24 Hours
  The score is rated on a scale from 0 to 10, where 0 indicates no pain and 10 indicates unbearable pain.